CLINICAL TRIAL: NCT03424304
Title: Open-label, Prospective, Single-Center Feasibility Study to Evaluate the Cutera Excel V™ Laser With Green Genesis and a Micro-Lens Array Attachment as Compared to the Standard-of-care With an Excel V™ Laser
Brief Title: Evaluation of Cutera Excel V™ Laser With Green Genesis and Micro-Lens Array (MLA)Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-17-EV12
Record Dates: First submitted 2017-12-13; First posted 2018-02-07 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Wrinkle; Rosacea; Scarring
MeSH Terms: conditions — Rosacea; Cicatrix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Excel V™ Laser With Green Genesis (Other): Treatment with Excel V™ Laser With Green Genesis and Micro-Lens Array (MLA)Attachment for skin quality in desired area
  Interventions: Device: Excel V™ Laser With Green Genesis

INTERVENTIONS:
Device: Excel V™ Laser With Green Genesis — Subject(s) will receive treatments with a Cutera Excel V™ Laser

SUMMARY:
Evaluate the Cutera excel V™ Laser with Green Genesis and a Micro-Lens Array (MLA) Attachment

DETAILED DESCRIPTION:
This is an open-label, prospective, single-center, split-face Feasibility study to Evaluate 1) the safety and efficacy of the Cutera excel V™ laser and the Micro-Lens Array attachment to the Genesis V hand piece, and 2) the safety and efficacy of the Cutera excel V™ laser Green Genesis V hand piece to the CoolView hand piece.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign the Informed Consent Form.
2. Female or Male, 18 to 65 years of age (inclusive).
3. Fitzpatrick Skin Type I - VI (Appendix 4).
4. Must be willing to have Cutera excel V laser treatments with MLA and/or Green Genesis (532 nm) and able to adhere to the treatments, follow-up visit schedule, and post-treatment care instructions.
5. Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.
6. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation (educational and/or marketing), publications, and any additional marketing purposes.
7. Agree to not undergo any other cosmetic procedure(s) or treatment(s) on the face during the study and has no intention of having such procedures performed during the course of the study.
8. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

1. Participation in a clinical trial of another drug, or device administered to the treatment area, within 3 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 3 months of study participation, such as laser procedures, facial fillers, toxins and those used for general aesthetic correction.
3. Use of prescription topicals in the treatment area within one month prior to treatment or use of topical agents one week prior to treatment that may cause facial sensitivity.
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
5. Pregnant and/or breastfeeding, or planning to become pregnant.
6. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.
7. Hypersensitivity to light exposure.
8. Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.
9. History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.
10. Has a history of squamous cell carcinoma or melanoma in the treatment area.
11. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
12. A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.
13. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
14. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
15. History of pigmentary disorders, particularly tendency for hyper- or hypo- pigmentation, or any that are considered not acceptable by the study investigator.
16. Has used oral isotretinoin (Accutane or therapeutic vitamin A supplements of equal to, or greater than 10,000 units per day) within 12 months of initial treatment or plans on using during the course of the study (note: skin must regain its normal degree of moisture prior to treatment, e.g. lack of noticeable skin flaking and peeling).
17. Excessively tanned or active sun tan in facial area to be treated, or unable/unlikely to refrain from tanning during the study.
18. Excessive facial hair in the area to be treated (beards, sideburns, and/or moustache,) that would interfere with diagnosis, assessment, and treatment.
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Cutera Research Center
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Excel V™ Laser With Green Genesis: Treatment with Excel V™ Laser With Green Genesis and Micro-Lens Array (MLA)Attachment
Period: Overall Study
Arm/Group | Excel V™ Laser With Green Genesis
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Excel V™ Laser With Green Genesis
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Global Aesthetic Improvement Scale
Description: The improvement after treatment on the Global Aesthetic Improvement Scale (GAIS).
  Higher scores mean better outcomes 4=Very Significant Improvement 3=Significant Improvement 2=Moderate Improvement
  1=Mild Improvement 0=No Change
Time Frame: 12 weeks post-final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Excel V™ Laser With Green Genesis
Number analyzed (Participants) | 19
score on a scale
  Right side of the face | 0.95 (1.40)
  Left side of the face | 1.05 (1.28)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks post-final treatment
Arm/Group | Excel V™ Laser With Green Genesis
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Excel V™ Laser With Green Genesis (N=20)
Erythema (Skin and subcutaneous tissue disorders) | 20
Edema (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT03424304/Prot_SAP_000.pdf